CLINICAL TRIAL: NCT04342546
Title: Prospective Evaluation of a Predictive Toxicity Test Post Radiotherapy After Mastectomy With Immediate Implant Reconstruction
Brief Title: Predictive Toxicity Test Linked to Radiotherapy After Mastectomy and Immediate Implant Reconstruction
Acronym: PRETORIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2019-07 PRE; 2019-A02178-49 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2020-03-25; First posted 2020-04-13 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Capsular Contracture Associated With Breast Implant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: For all the patients, the NovaGray RILA Breast® test will be performed between day -30 and until the first day of radiotherapy (before the start of this one) and then 12 months after the end of radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toxicity test (Experimental): For all patients, the NovaGray RILA Breast® test will be performed between day -30 and until the first day of radiotherapy (before the start of this one) and then 12 months after the end of radiotherapy and in the case of neoadjuvant chemotherapy, between day -30 and until the first day of chemotherapy (before any injection) and in the case of adjuvant chemotherapy, between day -30 and until the first day of chemotherapy (before any injection).
  The test consists of a blood sample of 2x4 mL
  Interventions: Device: NovaGray RILA Breast® test

INTERVENTIONS:
Device: NovaGray RILA Breast® test — The test consists of a blood sample of 2x4 mL. This test will be performed between day -30 and until the first day of radiotherapy (before the start of this one) and then 12 months after the end of radiotherapy and between day -30 and until the first day of chemotherapy (before any injection) in the case of neoadjuvant chemotherapy and between day -30 and until the first day of chemotherapy (before any injection) in the case of adjuvant chemotherapy.

SUMMARY:
This study evaluates the capacity of the NovaGray RILA Breast® test to predict the toxicity linked to radiotherapy and the impact of implant breast reconstruction.

DETAILED DESCRIPTION:
Immediate reconstruction after mastectomy may help women with breast cancer to deal with their fear of mastectomy, spare them one or more second surgery and additional hospital stays in case of late breast reconstruction. However, in France, most patients with invasive breast carcinoma and treated with mastectomy are not offered immediate reconstruction. One reason is the need for postoperative radiotherapy for most patients (40 to 70% according to the centers). Indeed, radiotherapy induces side-effects which can alter the cosmetic result of the breast reconstruction as well as the patient's quality of life. Since 1995, a significant correlation is observed between the RILA test (measurement by flux cytometry of the lymphocyte T-CD8 apoptosis induced by radiotherapy) and the risk of occurrence of severe radio-induced breast fibrosis. Such accurate personalized medical care could allow identifying before any treatment high risk of toxicity patients and thus help establishing the therapeutic strategy. Identification of low-risk patients could also allow limiting autologous samplings and thus their associated morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with histologically confirmed breast cancer with indication of mastectomy or surgery with mastectomy performed
* Indication of wall chest radiation after mastectomy
* Patient's agreement to receive or having had an immediate breast reconstruction by implant in one or two steps, with or without a dermal or synthetic matrix (depending on the habits of the center)
* Performance Status 0-1
* Consent signed before any study procedure
* Patient geographically accessible for follow-up
* Affiliated to the French national social security system

Exclusion Criteria:

* Breast reconstruction with flap
* Inflammatory breast cancer (cT4d)
* Skin or parietal breast cancer (cT4 a, b or c)
* Metastatic patients
* Patients with bilateral breast cancer
* History of homolateral breast cancer treated with radiotherapy
* History of contralateral breast cancer
* Pregnant or breastfeeding women
* Legal incapacity or physical, psychological or mental status interfering with the patient's ability to sign the informed consent
* Participation in an interventional clinical study or planned participation during study up to 12 months post-radiotherapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients with breast cancer treated by mastectomy with immediate implant breast reconstruction
Enrollment: 250 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Ability of a radiosensitivity test to predict capsular contracture | 12 months after the end of radiotherapy
  To identify the Area Under the Curve (AUC) of the radiosensitive predictive test of Grade 3-4 capsular contracture

SECONDARY OUTCOMES:
Capsular contracture prevalence | 12 Months
  Rate of capsular contracture after radiotherapy
Accuracy of the dichotomized test based on the optimal threshold | 12 months
  Accuracy of the test assessed by Sensitivity, Specificity, Positive Predictive Value and Negative Predictive Value
Precision of the radiosensitivity predictive test | 12 months
  Using the time dependant AUC (AUCt) method
Biological prognostics factors for capsular contracture occurence | 12 months
  Number and type of different biological prognostic factors of capsular contracture occurence
Tumoral prognostics factors for capsular contracture occurence | 12 months
  Number and type of different tumoral prognostic factors of capsular contracture occurence
Success of each surgical strategy in terms of deposit | 24 months
  Number of deposit according to each reconstruction surgery (one or two step)
Cosmetic outcomes measure | 6, 12, 18 and 24 months
  Cosmetic questionnaire : BREAST-Q
Functional outcomes measure | 6, 12, 18 and 24 months
  Functional questionnaire: BREAST-Q
Patient satisfaction measure | 6, 12, 18 and 24 months
  Patient satisfaction questionnaire: BREAST-Q
General quality of life measure | 6, 12, 18 and 24 months
  Quality of life questionnaire: QLQ-C30
Specific quality of life measure for breast cancer patient | 6, 12, 18 and 24 months
  Quality of life questionnaire for breast cancer patient: QLQ-BR23
Stability of the test after chemotherapy | 12 months
  Test score at 12 months after the end of radiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Marian Gutowski, Study Chair — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (9):
- France (9):
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - centre Antoine Lacassagne, Nice
  - Hôpital Tenon, Paris
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Negre G, Balcaen T, Dast S, Sinna R, Chazard E. Breast reconstruction in France, observational study of 140,904 cases of mastectomy for breast cancer. Ann Chir Plast Esthet. 2020 Feb;65(1):36-43. doi: 10.1016/j.anplas.2019.07.014. Epub 2019 Aug 2. PMID 31383624
- [Background] Ng SK, Hare RM, Kuang RJ, Smith KM, Brown BJ, Hunter-Smith DJ. Breast Reconstruction Post Mastectomy: Patient Satisfaction and Decision Making. Ann Plast Surg. 2016 Jun;76(6):640-4. doi: 10.1097/SAP.0000000000000242. PMID 25003439
- [Background] Howes BH, Watson DI, Xu C, Fosh B, Canepa M, Dean NR. Quality of life following total mastectomy with and without reconstruction versus breast-conserving surgery for breast cancer: A case-controlled cohort study. J Plast Reconstr Aesthet Surg. 2016 Sep;69(9):1184-91. doi: 10.1016/j.bjps.2016.06.004. Epub 2016 Jun 18. PMID 27406255
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Background] Ricci JA, Epstein S, Momoh AO, Lin SJ, Singhal D, Lee BT. A meta-analysis of implant-based breast reconstruction and timing of adjuvant radiation therapy. J Surg Res. 2017 Oct;218:108-116. doi: 10.1016/j.jss.2017.05.072. Epub 2017 Jun 15. PMID 28985836
- [Result] Barry M, Kell MR. Radiotherapy and breast reconstruction: a meta-analysis. Breast Cancer Res Treat. 2011 May;127(1):15-22. doi: 10.1007/s10549-011-1401-x. Epub 2011 Feb 20. PMID 21336948